CLINICAL TRIAL: NCT05642546
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of a Single Dose of NM8074 Administered Intravenously to Healthy Subjects
Brief Title: First-in-Human (FIH) Clinical Study of NM8074 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NovelMed Therapeutics (Industry)
Collaborators: Labcorp Corporation of America Holdings, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 06-101-FIH-NM8074
Record Dates: First submitted 2022-11-18; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-11

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Eligible subjects who meet the inclusion/exclusion criteria will be randomized on Day 1 to either NM8074 or placebo. The sentinel pair in each of the 5 dose cohorts will be randomized in a 1:1 ratio to receive NM8074 or placebo. The remaining subjects will be randomized in a 5:1 ratio to NM8074 to placebo. Dose escalation will occur in sequential cohorts once safety has been evaluated in the prior cohort.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study (subjects and on-site medical/nursing staff at the study site are blinded to study drug/dose assignment). The pharmacy staff preparing the investigational products will not be blinded to NM8074 study drug assignment, but all other site staff, including the Investigator, will be blinded. Unblinding should only be considered for the safety of the subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NM8074 (Experimental): 6 subjects per each of the 5 cohorts will receive a single dose of NM8074 administered via IV (intravenous) infusion at 0.3, 1.0, 3.0, 10, or 20 mg/kg
  Interventions: Drug: NM8074
- Placebo (Placebo Comparator): 2 subjects per each of the 5 cohorts will receive saline placebo administered via IV infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NM8074 — Novel, recombinant, humanized monoclonal antibody that selectively binds to human Factor Bb with high affinity and blocks the formation of Alternative Pathway (AP) driven C3 and C5 convertases
  Arms: NM8074
Drug: Placebo — Saline Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 1 randomized, double-blind, placebo-controlled, single administration, sequential cohort with sentinel dosing, dose escalation study designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and immunogenicity of NM8074 in healthy subjects. This study will include 5 cohorts, with each cohort consisting of a total of 8 healthy subjects, including both males and females, randomized in a 3:1 ratio of NM8074 to placebo (6 subjects assigned to NM8074 and 2 subjects assigned to placebo).

DETAILED DESCRIPTION:
NM8074 is a novel, recombinant, humanized monoclonal antibody. NM8074 selectively binds to human Factor Bb with high affinity and blocks the formation of Alternative Pathway (AP) driven C3 and C5 convertases. Both C3 and C5 convertases are critical for exacerbation and amplification of the AP in complement-mediated disorders. 06-101-FIH-NM8074 is the first-in-human clinical trial for NM8074 which is intended to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and immunogenicity of NM8074 when delivered as a single intravenous infusion to healthy volunteers. Doses will be escalated in each of the 5 sequential cohorts using sentinel dosing.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female subjects ≥18 years to ≤60 years of age, inclusive
* Body mass index (BMI) between 18 kg/m2 and 32 kg/m2, inclusive and weigh at least 50 kg
* QT interval (Fridericia's correction [QTcF]); QTcF ≤ 450 msec for males and ≤ 470 msec for females at Screening and prior to dosing on Admittance Day -1
* Willing and able to give signed Informed Consent and comply with the study visit schedule
* In good general health as determined by the Investigator's review of medical history, concomitant medications, physical examination, clinical laboratory tests, and ECG evaluations
* Male subjects must agree to use barrier contraception (male condom) and not donate sperm during the treatment period and for at least 3 months after the last dose of NM8074. Barrier contraception is required even with documented medical assessment of the surgical success of a vasectomy
* Female subjects who are of childbearing potential must use highly effective contraception1 or acceptable contraception as defined below, starting at screening and continuing until at least 3 months after the last dose of NM8074. Female subjects must not donate ova during the screening and treatment periods and for at least 3 months after the last dose of NM8074

Highly effective contraceptive methods for female subjects are as follows:

a. Combined (estrogen and progesterone containing) hormonal contraception associated with inhibition of ovulation: i. Oral contraceptives (e.g., oral, injected, implanted) or intrauterine ii. Intravaginal iii. Transdermal b. Progesterone-only hormonal contraception associated with inhibition of ovulation: i. Oral ii. Injectable iii. Implantable c. Intrauterine Device d. Intrauterine hormone-releasing system e. Bilateral tubal occlusion/tubal ligation (or comparable procedure)

* Women of Non-childbearing Potential

  a. Postmenopausal: i. 12 continuous months of natural (spontaneous) amenorrhea without an alternative medical cause and a serum follicle-stimulating hormone (FSH) level
  * 40 mIU/mL ii. 6 weeks after surgical bilateral oophorectomy with or without hysterectomy b. Post-hysterectomy
* Sexual Abstinence Subjects who practice true abstinence, because of the subject's lifestyle choice (i.e., the subject should not become abstinent just for the purpose of study participation), are exempt from contraceptive requirements. Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception. For subjects who practice true abstinence, subjects must be abstinent for at least 6 months prior to screening and must agree to remain abstinent from the time of signing the Informed Consent Form until the end of study.
* Same-sex Relationships For subjects who are exclusively in same-sex relationships, contraceptive requirements do not apply. A subject in a same-sex relationship at the time of signing the Informed Consent Form (ICF) must agree to refrain from engaging in a heterosexual relationship from the time of signing the ICF until the end of study
* Has received the MenB Bexsero® vaccination against Neisseria meningitidis serogroup B (consisting of 2 intramuscular injections, 30 days apart) with the first injection at least 45 days prior to study drug initiation, and the second injection no later than 15 days prior to study drug initiation, and/or provides documentation of positive titer response precluding revaccination
* Has received the MenACWY Menactra® polysaccharide diphtheria toxoid conjugate vaccine solution against Neisseria meningitidis serogroups A, C, Y, and W-135 (consisting of 1 intramuscular injection) at least 45 days prior to study drug initiation with confirmation of response acceptable by PI, and/or provides documentation of positive titer response precluding re-vaccination
* Negative serum pregnancy test at Screening and Check-In for all female subjects
* Only non-smokers will take priority in enrollment for the study. Should there be a shortage of available healthy volunteers, light smokers (~10 cigarettes/day) will be accepted

Exclusion Criteria:

* Subjects who plan to travel during the course of the study to endemic areas as per the Centers for Disease Control and Prevention (CDC) definition for meningococcal meningitis
* Has a currently active systemic infection that requires antibiotic, antifungal, antiparasitic, or antiviral medications. Any infection prior to entry into the study must have been cured for 1 month prior to the Screening Visit
* Positive QuantiFERON®-TB test indicating possible tuberculosis (TB) infection, active systemic bacterial, viral, or fungal infection within 14 days prior to dosing
* Has a known history of meningococcal/pneumococcal/gonococcal disease
* Contraindication to receiving meningococcal vaccine, including severe (life-threatening) allergic reaction to a previous dose of meningococcal serogroup B vaccine; severe (life-threatening) allergy to any vaccine component; previous diagnosis of Guillain-Barré Syndrome
* History of unexplained, recurrent infection; or infection requiring treatment with systemic antibiotics within the last 90 days prior to dosing
* History of latent or active tuberculosis or exposure to endemic areas within 8 weeks prior to the tuberculosis test performed at screening
* Clinically significant abnormalities in urine upon urinalysis to allow investigator discretion and to prevent disqualifications for minor findings of no significance such as mucus in the urine
* Any of the following hematology tests: hemoglobin; total white blood cells (total WBC); absolute neutrophils; and platelets outside the laboratory reference range at Screening and Day -1
* Abnormal urine tests: Clinically significant abnormalities in urine upon urinalysis" to allow investigator discretion and to prevent disqualifications for minor findings of no significance such as mucus in the urine
* History of continuous topical/inhaled or systemic steroid use > 1 month or history of any inhaled or topical immunosuppressive therapy within 90 days prior to study drug administration
* Has any history of or active cardiac disease, including congestive heart failure, angina, any arrhythmia, or clinically significant findings on ECGs
* Has asthma or other severe respiratory disease (e.g., chronic obstructive pulmonary disease) requiring daily prescription medication or prior emergency room visits or hospitalization
* Has a history of solid organ transplantation; or has kidney, neurologic, metabolic, or other organ system disease that, in the Investigator's opinion, precludes participation in this study
* Has clinically significant liver disease or transaminase (alanine aminotransferase [ALT] and aspartate aminotransferase [AST] levels > 1.5x the upper limit of normal (ULN) measured at Screening and Day-1
* Has total bilirubin levels > 1.5x ULN measured at Screening
* Has an estimated glomerular filtration rate <70 mL/minute/1.73m2 measured at Screening (measured with creatinine clearance or Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI))
* Has an abnormal laboratory finding or vital signs outside the specified normal parameters at the Screening Visit which is judged by the PI as clinically significant
* Has any clinically significant ECG abnormality at Screening or Check-In
* History of allergy to excipients of NM8074
* Use of prescription medications within 28 days prior to study drug administration
* Has a body temperature >99.5 °F (37.5 °C) a fever associated with a symptomatic viral or bacterial infection) within 2 weeks prior to the first dosing
* Has an immunological disorder such as, but not limited to, human immunodeficiency virus (HIV); acquired or congenital immune deficiency syndrome; autoimmune diseases, such as, but not limited to, rheumatoid arthritis, systemic lupus erythematosus, vasculitis, or seronegative spondyloarthropathies; or any acute or chronic infection, including, but not limited to, hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Is pregnant, lactating, or planning a pregnancy
* Has used any prescribed medication within 14 days prior to the first admission or has plans to use any prescribed medication during the study (with the exception of hormonal contraceptives)
* Participation in any experimental small molecule or non-antibody molecule therapy within 60 days prior to dosing on Day 1
* Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at Screening) of more than 50 mL of blood within 30 days of dosing, or more than 499 mL of blood within 56 days of dosing
* Immunization with a live attenuated vaccine 1 month prior to dosing or planned vaccination during the course of the study (except for the vaccination planned by the study protocol)
* History of use of illegal recreational drugs within 1 year prior to Screening
* Has used any over-the-counter medicinal products, including herbal and dietary supplements, within 7 days prior to the first admission or has plans to use during the study (with the exception of approved daily doses of acetaminophen, ibuprofen, or aspirin for the treatment of minor discomfort)
* Is currently participating in any other type of clinical trial
* Has previously been randomized and withdrawn from this study
* Has active alcohol or substance abuse or history of alcohol or substance abuse within the 6 months prior to randomization or has a positive result on urine drug or breath alcohol screen during the Screening Visit. The use of alcohol is prohibited for 48 hours prior to Check-In and during confinement.
* Subjects with any medical history, conditions, or risks, which, in the opinion of the Investigator, may interfere with the subject's full participation in the study, or compliance with the protocol, poses any additional risk for the subject, or confounds the assessment of the subject or outcome of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Monitoring of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 71 days post-dose
  Adverse events will be graded according to the CTCAE v4.03. If the AE term is not described in the grading scales, the AE severity shall be reported according to the following:
  * Grade I: Mild (awareness of sign or symptom, but easily tolerated)
  * Grade II: Moderate (discomfort sufficient to cause interference with normal activities)
  * Grade III: Severe (incapacitating, with inability to perform normal activities)
  * Grade IV: Life threatening
  * Grade V: Fatal

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) | Up to 71 days post-dose
Time to maximum observed serum concentration (tmax) | Up to 71 days post-dose
Area under the serum concentration versus time curve from time zero to the last quantifiable concentration (AUCt) | Up to 71 days post-dose
AUC from time zero to infinity (AUC∞) | Up to 71 days post-dose
Terminal elimination rate constant (λz) | Up to 71 days post-dose
Terminal half-life (t½) | Up to 71 days post-dose
Total clearance (CL) | Up to 71 days post-dose
Volume of distribution (Vd) | Up to 71 days post-dose
Change from Baseline or Percent Change from Baseline in Levels of Complement Component C3b via Alternative Pathway (AP) of Complement Activity | Up to 71 days post-dose
Change from Baseline or Percent Change from Baseline in Levels of Membrane Attack Complex (MAC) via the Alternative Pathway (AP) of Complement Activity | Up to 71 days post-dose
Number of Participants with Antidrug Antibodies (ADAs) to NM8074 | Up to 71 days post-dose

OTHER OUTCOMES:
Change from Baseline or Percent Change from Baseline in Complement Component Factor B | Up to 71 days post-dose
Change from Baseline or Percent Change from Baseline in Levels of Membrane Attack Complex via Classical Pathway (CP) of Complement Activity | Up to 71 days post-dose
Change from Baseline or Percent Change from Baseline in Levels of Complement Component C3b via Classical Pathway (CP) of Complement Activity | Up to 71 days post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Unit, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No